CLINICAL TRIAL: NCT03466047
Title: A Physiological Study on the Effect of Macronutrients Delivery to the Proximal and Distal Small Bowel on Satiety and Gut Hormone Responses
Brief Title: The Effect of Macronutrients on Satiety and Gut Hormone Responses
Acronym: Microcapsule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Carel Le Roux, Professor, Imperial College London
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Microcapsule
Record Dates: First submitted 2018-03-03; First posted 2018-03-15 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Protein stomach (Experimental): Encapsulated protein released in the stomach
  Interventions: Dietary Supplement: Protein stomach
- Protein distal small intestine (Experimental): Encapsulated protein released in the distal small intestine
  Interventions: Dietary Supplement: Protein distal small intestine
- CHO stomach (Experimental): Encapsulated CHO released in the stomach
  Interventions: Dietary Supplement: CHO stomach
- CHO distal small intestine (Experimental): Encapsulated CHO released in the distal small intestine
  Interventions: Dietary Supplement: CHO distal small intestine
- Fat stomach (Experimental): Encapsulated Fat released in the stomach
  Interventions: Dietary Supplement: Fat stomach
- Fat distal small intestine (Experimental): Encapsulated Fat released in the distal small intestine
  Interventions: Dietary Supplement: Fat distal small intestine

INTERVENTIONS:
Dietary Supplement: Protein stomach — encapsulated protein stomach
  Arms: Protein stomach
Dietary Supplement: Protein distal small intestine — encapsulated protein distal small intestine
  Arms: Protein distal small intestine
Dietary Supplement: CHO stomach — encapsulated CHO stomach
  Arms: CHO stomach
Dietary Supplement: CHO distal small intestine — encapsulated CHO distal small intestine
  Arms: CHO distal small intestine
Dietary Supplement: Fat stomach — encapsulated Fat stomach
  Arms: Fat stomach
Dietary Supplement: Fat distal small intestine — encapsulated Fat distal small intestine
  Arms: Fat distal small intestine

SUMMARY:
This study is part of a research theme aiming at elucidating the physiological mechanisms of action of weight loss after gastric bypass surgery. The Roux-en-Y Gastric Bypass procedure induces pronounced and sustained weight loss, but the physiological mechanisms of action are not completely clear. Neither mechanical restriction of food intake nor malabsorption, are the main contributing factors. The enhanced postprandial responses of gut hormones (e.g. GLP-1 and PYY) which increase satiety as well as energy expenditure after surgery suggest a changed physiological set point for appetite and metabolism.

Our hypothesis is that the intake of high quantity of protein in a microcapsule form would be able to reach the distal parts of the intestinal mucosa and stimulate maximum stimulation of the anorectic gut hormones. The higher functions of the brain will respond to these strong neuroendocrine signals by ensuing satiety and fullness.

DETAILED DESCRIPTION:
Ten healthy volunteers, aged 18 to 65 years will be recruited. Each subject will be studied on six occasions one week apart. On each visit, a baseline serum sample will be drawn from each subject. In a randomized way all subjects will receive the following meals in their successive weekly visits: Option 1 High protein mixed meal in capsules that break down in the stomach, Option 2 High protein mixed meal in capsules that break down in the distal small bowel, Option 3 High fat mixed meal in capsules that break down in the stomach, Option 4 High fat mixed meal in capsules that break down in the distal small bowel, Option 5 High CHD mixed meal in capsules that break down in the stomach, Option 6 High CHD mixed meal in capsules that break down in the distal small bowel. On the same day, all subjects will be offered standard ad libitum meal to measure their food consumption. After 3 hours (i.e. at 12:00) another blood sample will be drawn. All subjects will be asked to rate their appetite on a Visual Analogue Scale (VAS). Upon VAS completion the subjects will be allowed to go home.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Normal fasting glucose
* Stable body weight for at least last three months
* BMI < 30 Kg/m2
* Capacity to consent to participate
* Independently mobile

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded:
* Pre-diabetes Diabetes
* Obesity
* Smoking
* Substance abuse
* Pregnancy
* Use of medications (except for oral contraceptives)
* Chronic medical or psychiatric illness
* Any significant abnormalities detected on physical examination, electrocardiography, or screening blood tests (measurement of complete blood count, electrolytes, fasting glucose, and liver function)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carel le Roux, Principal Investigator — Imperial College London
Locations (1):
- Clinical Research Centre, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Interventions: 6 interventions
Period: Protein Stomach (1day)
Arm/Group | Interventions
Started | 8 (The same 8 patients were studied in all interventions)
Completed | 8 (The same 8 patients were studied in all interventions)
Not Completed | 0
Period: Protein Small Intestine (1 Day)
Arm/Group | Interventions
Started | 8
Completed | 8
Not Completed | 0
Period: CHO Stomach (1 Day)
Arm/Group | Interventions
Started | 8
Completed | 8
Not Completed | 0
Period: CHO Small Intestine (1 Day)
Arm/Group | Interventions
Started | 8
Completed | 8
Not Completed | 0
Period: Fat Stomach (1 Day)
Arm/Group | Interventions
Started | 8
Completed | 8
Not Completed | 0
Period: Fat Small Intestine (1 Day)
Arm/Group | Interventions
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Interventions: Encapsulated macronutrients in a drink, 6 experiments, Protein released in the stomach (1 day), Protein released in the small intestine (1 day), CHO released in the stomach (1 day), CHO released in the small intestine (1 day), Fat released in the stomach (1 day), fat released in the small intestine (1 day).
Arm/Group | Interventions
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (3.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Women | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 8
Weight [Mean (Standard Deviation); unit: kg] | 81.8 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Proteins on the Secretion of Gut Hormones From Different Parts of the Gastrointestinal Tract
Description: 3 hours AUC for different gut hormones (PYY) to determine the response to macronutrients in different release (stomach vs small intestine) locations. AUC for timepoints 0, 30min, 60min, 120min, 180min.
Time Frame: 3 hours
Measure: Mean (Standard Error); unit: pg*min/mL
Groups:
- Protein Stomach; Fat Stomach; CHO Stomach; Protein Distal Small Intestine; Fat Distal Small Intestine; CHO Distal Small Intestine: encapsulated protein made up into a flavored water drink
  A single macronutrient captured in microcapsules: Encapsulated macronutrients in a drink
Arm/Group | Protein Stomach | Fat Stomach | CHO Stomach | Protein Distal Small Intestine | Fat Distal Small Intestine | CHO Distal Small Intestine
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
pg*min/mL | 1310 (102) | 1073 (154) | 1118 (150) | 1188 (121) | 1725 (351) | 1194 (221)

2. Secondary Outcome: Total Intake (kj) of ad Libitum Lunch Meals to Assess Food Intake
Description: Food intake as assessed with ad libitum lunch 3 hours after intervention
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: kj
Arm/Group | Protein Stomach | Protein Distal Small Intestine | CHO Stomach | CHO Distal Small Intestine | Fat Stomach | Fat Distal Small Intestine
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
kj | 3138 (175) | 3389 (161) | 3146 (168) | 3008 (192) | 3690 (170) | 2305 (183)

3. Secondary Outcome: Visual Analogue Scale Ratings of Hunger
Description: Visual Analogue Scale ratings of hunger at 180 min (before the meal). The scale is 10cm line with two anchors at each end. Scores are recorded by making a handwritten mark that represents a continuum between "not hungry at all" and "Extremly hungry."
  The score of 0 represents least hunger. The score of 10 represent extreme hunger.
Time Frame: 180min
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Protein Small Intestine: Encapsulated protein released in small intestine
- CHO Stomach: CHO released in the stomach
- CHO Small Intestine: Encapsulated CHO released in the small intestine
- Fat Small Intestine: Encapsulated fat released in the small intestine
Arm/Group | Protein Stomach | Protein Small Intestine | CHO Stomach | CHO Small Intestine | Fat Stomach | Fat Small Intestine
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
cm | 5.4 (0.5) | 5.5 (0.5) | 3.8 (0.7) | 4.1 (0.6) | 4.1 (0.4) | 4.1 (0.5)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Protein Stomach | Fat Stomach | CHO Stomach | Protein Distal Small Intestine | Fat Distal Small Intestine | CHO Distal Small Intestine
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protein Stomach (N=8) | Fat Stomach (N=8) | CHO Stomach (N=8) | Protein Distal Small Intestine (N=8) | Fat Distal Small Intestine (N=8) | CHO Distal Small Intestine (N=8)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Loose Stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT03466047/Prot_SAP_000.pdf